CLINICAL TRIAL: NCT04087122
Title: Evaluate the Efficiency Impact of Conducting Active Temperature Management During Cardiac Cryoablation Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Cooling Therapy, Inc., d/b/a Attune Medical (Industry)
Collaborators: Winchester Medical Center (Other)
Responsible Party: Sponsor
Organization: Advanced Cooling Therapy LLC, d/b/a Attune Medical (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WMC-Cryo
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Esophageal warming (Experimental): Patients receive the Attune Medical Esophageal Heat Transfer Device
  Interventions: Device: Esophageal warming device (Attune Medical, Chicago, IL

INTERVENTIONS:
Device: Esophageal warming device (Attune Medical, Chicago, IL — Prospective, single center pilot stud

SUMMARY:
Left atrial catheter ablation including pulmonary vein isolation is a standard therapy in the management of symptomatic atrial fibrillation; however thermal esophageal injury is a known potential consequence of this procedure. Delivery of radiofrequency (RF) energy necessary to perform left atrial ablation has the potential to cause injury to the nearby esophagus including ulceration, hematoma, spasm, esophageal motility disorders, and, in the most extreme case, atrial-esophageal fistula.Esophageal mucosal lesions are the likely precursor to AEF, and esophageal mucosal lesions have been detected on post-ablation endoscopy after pulmonary vein isolation with an incidence ranging from 3% to 60%.

Active esophageal cooling during RF ablation as a means of esophageal injury prevention has been investigated through mathematical models, pre-clinical studies, and in clinical trials. Existing data support the efficacy of this approach, but the practice has not been widely adopted due to lack of a commercially available device.

The aim of this study is to evaluate the impact on procedural efficiency of ablation procedures performed using esophageal heat transfer to warm the esophagus during left atrial cryoablation.

DETAILED DESCRIPTION:
This study is a prospective, pilot study using the Attune Medical ensoETM esophageal heat transfer device to actively warm the esophagus during cryoablation procedures. This design is appropriate to gather the data needed regarding overall procedural time, compare this to historical controls, and estimate a sample size for a larger study powered for statistical significance.

Once patient consent is obtained, the subject will undergo preparation and anesthesia procedures following standard practice. Once the patient is intubated, the esophageal heat transfer device will be placed into the esophagus according to the IFU. The device will remain in place until the ablation procedure is completed and will be removed before extubation. Left atrial cryoablation using the standard approach will be performed with the ensoETM set at a temperature of 42 degrees C.

All patients will be followed up in total for 6 weeks (Long Term FU visit) after the procedure to document any clinical complication related to thermal esophageal injuries if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age over 18 years).
* Undergoing cryoablation for the treatment of atrial fibrillation, including pulmonary vein isolation.
* Patients must be able to understand and critically review the informed consent form.
* Subjects must understand and agree to study requirements and sign a written informed consent.

Exclusion Criteria:

* Patients who are unable to provide informed consent.
* Significant co-morbidities that preclude standard ablation procedure.
* Patients with <40 kg of body mass.
* Patients with relevant esophageal pathology (e.g. esophageal cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Alexander, MD, Principal Investigator — Winchester Medical Center; Zachary Hollis, MD, Principal Investigator — Winchester Medical Center
Locations (1):
- Winchester Medical Center, Winchester, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Esophageal Warming
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Esophageal Warming
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Total Time of Active Ablation Procedure
Description: Total time of active ablation procedure measured from trans-septal puncture to achievement of Pulmonary Vein Isolation (PVI)
Time Frame: Study Day 1 for all patients enrolled, during left atrial ablation procedures using cryoablation
Measure: Mean (95% Confidence Interval); unit: minutes
Groups:
- Esophageal Warming: Patients receiving the Attune Medical Esophageal Heat Transfer Device
Arm/Group | Esophageal Warming
Number analyzed (Participants) | 20
minutes | 126 [112 to 139]

2. Secondary Outcome: Total Procedure Time
Description: Total procedure time from patient entry to Electrophysiology (EP) lab until discharge to Post-Anesthesia Care Unit (PACU)
Time Frame: Study Day 1 for all patients enrolled from patient entry to Electrophysiology (EP) lab until post procedure discharge to Post-Anesthesia Care Unit (PACU)]
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Esophageal Warming
Number analyzed (Participants) | 20
minutes | 126 [112 to 139]

3. Secondary Outcome: Number of Procedural Pauses During Left Atrial Instrumentation
Description: Number of procedural pauses during left atrial instrumentation measured from trans-septal puncture to achievement of Pulmonary Vein Isolation (PVI)
Time Frame: Study Day 1 for all patients, during left atrial ablation procedures using cryoablation
Measure: Mean (95% Confidence Interval); unit: Procedural pauses
Arm/Group | Esophageal Warming
Number analyzed (Participants) | 20
Procedural pauses | 0 [0 to 16.8]

4. Secondary Outcome: Total Duration of Fluoroscopy Use
Description: Total duration of fluoroscopy use during left atrial instrumentation measured from trans-septal puncture to achievement of Pulmonary Vein Isolation (PVI)
Time Frame: Study Day 1 for all patients, during left atrial ablation procedures using cryoablation
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Esophageal Warming
Number analyzed (Participants) | 20
minutes | 23.4 (7.8)

ADVERSE EVENTS:
Time Frame: 145 days
Description: All-Cause Mortality; Serious Adverse Events; Other (Not Including Serious) Adverse Events
Arm/Group | Esophageal Warming
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT04087122/Prot_SAP_000.pdf